CLINICAL TRIAL: NCT01871181
Title: The Short and Long-term Effects of Ultrasound-guided Ilioinguinal and Iliohypogastric Nerve Block on Postoperative Pain Control Following Open Inguinal Hernia Repair
Brief Title: US-guided Ilioinguinal Blocks Versus Local Infiltration
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer at institution
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00026522
Record Dates: First submitted 2013-06-03; First posted 2013-06-06 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2016-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ilioinguinal block (Experimental): Patients in this group will receive an ultrasound-guided ilioinguinal nerve block.
  Interventions: Procedure: Ilioinguinal block
- Local infiltration (Active Comparator): Patients in this group will receive the standard method of local infiltration of local anesthetic around the surgical site.
  Interventions: Procedure: Local infiltration

INTERVENTIONS:
Procedure: Ilioinguinal block — 0.25% bupivacaine will be administered on a mg/kg basis
  Arms: Ilioinguinal block
Procedure: Local infiltration — Surgeon will infiltrate incision area with local anesthetic before closure.
  Arms: Local infiltration

SUMMARY:
Injection of local anesthetic drugs is an effective way to freeze (block) nerves to achieve loss of sensation during surgery and satisfactory pain control afterwards. Many studies have shown that nerve block is associated with higher degree of success in controlling pain after open inguinal hernia repair. Nerve block can be administered by a single injection with a long acting local anesthetic agent using ultrasound guidance. This study is to compare different techniques for freezing the nerves responsible for pain after open inguinal hernia repair. Patients will be randomized to one of two groups. In the first group, participants will receive ultrasound-guided nerve block following induction of general anesthesia but prior to surgical procedure. In the second group, participants will receive local anesthetic injection directly into the wound by the surgeon prior to closure. The investigators will assess the level of pain control for 48 hours after the surgical procedure. Patients will be provided with additional medications for pain relief if necessary. The investigators will also contact participants to follow-up with regard to possible chronic groin pain after 3 months following the surgical procedure.

DETAILED DESCRIPTION:
populations. It is well-known that inguinal hernia surgery can lead to significant degree of acute perioperative pain. At the same time, patients undergoing inguinal hernia operation are at increased risk to develop chronic neuropathic groin pain. In the literature, several approaches to prophylaxis and treatment of perioperative pain have been described including: infiltration of local anesthetics by surgeons, ilioinguonal/iliohypogastric nerve blocks, neuroaxial blockade, and caudal block in pediatric petients.

Recent studies have shown that ultrasound guided ilioinguinal/iliohypogastric nerve block is associated with increased level of safety, improved success rate, and reduction in dose of local anesthetic required compared to the "blind" technique.

The aim of our study is to investigate the role of ultrasound guided ilioinguinal/iliohypogastric nerve block in prevention of perioperative and persistent neuropathic pain following open inguinal hernia repair in comparison with infiltration of local anesthetics by surgeons. In the first randomized group of patients we will perform ultrasound guided ilioinguinal/iliohypogastric nerve block using the same types and amount of local anesthetics. In the second group, patients will receive infiltration of the same type and amount of local anesthetics by surgeons.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* Both gender
* 18 years and older
* Informed consent

Exclusion Criteria:

* ASA 4 and more
* Lack of informed consent
* Patients with history of chronic pain
* Patients on regular opioids
* History of allergic reaction to local anesthetics
* Medication or non-medication induced bleeding diastasis
* Infection at the site of injection
* Patients with bilateral hernias
* linguistic difficulties

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 48 hours post-surgery
  Pain will be recorded on a VAS scale immediately following surgery and then 24 and 48 hours post-surgery.

SECONDARY OUTCOMES:
Chronic pain | 6 months post-surgery
  All patients will be interviewed 3 and 6 months following the surgery in our chronic pain clinic or on the phone to evaluate the incidence of chronic groin pain in both groups.
Analgesic consumption | 48 hours post-surgery
  Consumption of all opioidal and non-opioidal analgesics will be recorded during the 48-hour period after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Klaassen Z, Marshall E, Tubbs RS, Louis RG Jr, Wartmann CT, Loukas M. Anatomy of the ilioinguinal and iliohypogastric nerves with observations of their spinal nerve contributions. Clin Anat. 2011 May;24(4):454-61. doi: 10.1002/ca.21098. Epub 2011 Jan 3. PMID 21509811
- [Background] Ndiaye A, Diop M, Ndoye JM, Ndiaye A, Mane L, Nazarian S, Dia A. Emergence and distribution of the ilioinguinal nerve in the inguinal region: applications to the ilioinguinal anaesthetic block (about 100 dissections). Surg Radiol Anat. 2010 Jan;32(1):55-62. doi: 10.1007/s00276-009-0549-0. Epub 2009 Aug 26. PMID 19707710
- [Background] Andersen FH, Nielsen K, Kehlet H. Combined ilioinguinal blockade and local infiltration anaesthesia for groin hernia repair--a double-blind randomized study. Br J Anaesth. 2005 Apr;94(4):520-3. doi: 10.1093/bja/aei083. Epub 2005 Feb 4. PMID 15695545
- [Background] Jagannathan N, Sohn L, Sawardekar A, Ambrosy A, Hagerty J, Chin A, Barsness K, Suresh S. Unilateral groin surgery in children: will the addition of an ultrasound-guided ilioinguinal nerve block enhance the duration of analgesia of a single-shot caudal block? Paediatr Anaesth. 2009 Sep;19(9):892-8. doi: 10.1111/j.1460-9592.2009.03092.x. Epub 2009 Jul 13. PMID 19627532
- [Background] Suresh S, Patel A, Porfyris S, Ryee MY. Ultrasound-guided serial ilioinguinal nerve blocks for management of chronic groin pain secondary to ilioinguinal neuralgia in adolescents. Paediatr Anaesth. 2008 Aug;18(8):775-8. doi: 10.1111/j.1460-9592.2008.02596.x. PMID 18482237
- [Background] Wang H. Is ilioinguinal-iliohypogastric nerve block an underused anesthetic technique for inguinal herniorrhaphy? South Med J. 2006 Jan;99(1):15. doi: 10.1097/01.smj.0000197300.37083.a8. No abstract available. PMID 16466114
- [Background] Wehbe SA, Ghulmiyyah LM, Dominique el-KH, Hosford SL, Ehleben CM, Saltzman SL, Sills ES. Prospective randomized trial of iliohypogastric-ilioinguinal nerve block on post-operative morphine use after inpatient surgery of the female reproductive tract. J Negat Results Biomed. 2008 Nov 28;7:11. doi: 10.1186/1477-5751-7-11. PMID 19040739